CLINICAL TRIAL: NCT04958291
Title: A Phase 1 Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of CC 99677 in Healthy Adult Japanese Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CC-99677 in Healthy Adult Japanese Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-99677-CP-004
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; CC-99677; Phase 1; Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Administration of Dose A of CC-99677 or Placebo (Experimental): Administration of Dose A of CC-99677 or Placebo
  Interventions: Drug: CC-99677; Other: Placebo
- Administration of Dose B of CC-99677 or Placebo (Experimental): Administration of Dose B of CC-99677 or Placebo
  Interventions: Drug: CC-99677; Other: Placebo
- Administration of Dose C of CC-99677 or Placebo (Experimental): Administration of Dose C of CC-99677 or Placebo
  Interventions: Drug: CC-99677; Other: Placebo

INTERVENTIONS:
Drug: CC-99677 — CC-99677
Other: Placebo — Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and pharmacogenomics (PG) of multiple doses of CC-99677 in healthy Japanese adult participants. This study will be placebo-controlled to appropriately characterize the safety and tolerability of CC-99677.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Participant is ≥ 18 and ≤ 55 years of age at the time of signing the informed consent form (ICF).
2. Japanese participants must have both paternal and both maternal grandparents be ethnically Japanese.
3. Participants must adhere to protocol-specified contraception requirements.
4. Participant has a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
5. Participant has physical exam, vital signs, clinical laboratory safety and other medical test results that are within normal limits, considered not clinically significant by the Investigator, or within other parameters specified in the protocol.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Participant has any significant medical condition (including but not limited to neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
2. Participant has any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
3. Participant is pregnant or breastfeeding.
4. Participant was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
5. Participant has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days prior to the first dose administration. Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
6. Participant has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration. Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
7. Participant has used CYP3A inducers and/or inhibitors (including St. John's Wort) within 30 days preceding the first dose administration.
8. Participant has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, or excretion, e.g., bariatric procedure. Appendectomy and cholecystectomy are acceptable. Other previous surgeries may be acceptable with concurrence of the Sponsor's Medical Monitor.
9. Participant donated blood or serum within 8 weeks before the first dose administration to a blood bank or blood donation center.
10. Participant smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
11. Participant has received immunization with a live or live attenuated vaccine within 2 months prior to the first dose administration or is planning to receive immunization with a live or live attenuated vaccine for 2 months following the last dose administration.
12. Participant has a history of Gilbert's syndrome or has laboratory findings at screening that, in the opinion of the Investigator, are indicative of Gilbert's syndrome.
13. Participant has a history of incompletely treated Mycobacterium tuberculosis (TB) infection, or has a positive QuantiFERON®-TB Gold (or equivalent) test at screening or 2 successive indeterminate QuantiFERON®-TB Gold (or equivalent) tests at screening.
14. Participants with clinical symptoms or signs (including febrile illness) suggesting active, subacute, or unresolved chronic infection.
15. Previous SARS-CoV-2 infection within 4 weeks prior to screening.

    a. Symptoms must have completely resolved and, based on Investigator assessment in consultation with the Sponsor's Medical Monitor, there are no sequelae that would place the participant at a higher risk of receiving IP.
16. Participant has previously been exposed to CC-99677 (e.g., in a prior clinical trial).
17. Participant has a history of photosensitivity to medications.
18. Participant is part of the study site staff personnel or a family member of the study site staff.
19. Any other exclusion criteria specified in the protocol that will be made known to participants prior to signing ICF.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From enrollment until at least 28 days after last dose of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax for CC-99677 | Up to 48 hours after last dose of study treatment
  Maximum observed plasma concentration within a dosing interval
Pharmacokinetics - tmax for CC-99677 | Up to 48 hours after last dose of study treatment
  Time of maximum observed plasma concentration within a dosing interval
Pharmacokinetics - AUCtau for CC-99677 | Up to 48 hours after last dose of study treatment
  Area under the plasma concentration-time curve within a dosing interval
Pharmacokinetics - AUC0-ti for CC-99677 | Up to 48 hours after last dose of study treatment
  Area under the plasma concentration-time curve from time zero to time ti within a dosing interval
Pharmacokinetics - Ctau for CC-99677 | Up to 48 hours after last dose of study treatment
  Concentration at the end of a dosing interval
Pharmacokinetics - Ctrough for CC-99677 | Up to 48 hours after last dose of study treatment
  Trough observed plasma concentration
Pharmacokinetics - t½ for CC-99677 | Up to 48 hours after last dose of study treatment
  Apparent terminal phase half-life
Apparent terminal phase half-life | Up to 48 hours after last dose of study treatment
  Apparent total body clearance
Pharmacokinetics - Vz/F for CC-99677 | Up to 48 hours after last dose of study treatment
  Apparent volume of distribution of terminal phase
Pharmacokinetics - DF for CC-99677 | Up to 48 hours after last dose of study treatment
  Degree of fluctuation
Pharmacokinetics - Css-avg for CC-99677 | Up to 48 hours after last dose of study treatment
  Average concentration within a dosing interval
Pharmacokinetics - AI_Cmax for CC-99677 | Up to 48 hours after last dose of study treatment
  Ratio of Cmax at steady-state to Cmax after the first dose
Pharmacokinetics - AI_AUC for CC-99677 | Up to 48 hours after last dose of study treatment
  Ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose
Pharmacokinetics - Cmax for CC0782951 | Up to 48 hours after last dose of study treatment
  Maximum observed plasma concentration within a dosing interval
Pharmacokinetics - tmax for CC0782951 | Up to 48 hours after last dose of study treatment
  Time of maximum observed plasma concentration within a dosing interval
Pharmacokinetics - AUCtau for CC0782951 | Up to 48 hours after last dose of study treatment
  Area under the plasma concentration-time curve within a dosing interval
Pharmacokinetics - AUC0-ti for CC0782951 | Up to 48 hours after last dose of study treatment
  Area under the plasma concentration-time curve from time zero to time ti within a dosing interval
Pharmacokinetics - Ctau for CC0782951 | Up to 48 hours after last dose of study treatment
  Concentration at the end of a dosing interval
Pharmacokinetics - Ctrough for CC0782951 | Up to 48 hours after last dose of study treatment
  Trough observed plasma concentration
Pharmacokinetics - t½ for CC0782951 | Up to 48 hours after last dose of study treatment
  Apparent terminal phase half-life
Pharmacokinetics - DF for CC0782951 | Up to 48 hours after last dose of study treatment
  Degree of fluctuation
Pharmacokinetics - Css-avg for CC0782951 | Up to 48 hours after last dose of study treatment
  Average concentration within a dosing interval
Pharmacokinetics - AI_Cmax for CC0782951 | Up to 48 hours after last dose of study treatment
  Ratio of Cmax at steady-state to Cmax after the first dose
Pharmacokinetics - AI_AUC for CC0782951 | Up to 48 hours after last dose of study treatment
  Ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Local Institution - 001, Long Beach, California

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm